CLINICAL TRIAL: NCT05215457
Title: Severity Indices of Diquat Poisoning for Triage and Prognosis in Acute Diquat Poisoning: A Multicenter Prospective Cohort Study
Brief Title: Severity Indices of Diquat Poisoning for Triage and Prognosis in Acute Diquat Poisoning
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hao Sun, MD, PhD, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2021-SR-394
Record Dates: First submitted 2022-01-01; First posted 2022-01-31 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Diquat Poisoning
Keywords: diquat; poisoning; triage; prognosis; survival analysis
MeSH Terms: conditions — Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Development Set: The development set included 106 patients, comprising 67 survivors and 39 fatalities, with a case fatality rate of 36.8%; 56.6% were men. Data from the study center (teaching hospital affiliated to Nanjing Medical University) were used for model development.
- External Validation Set: The external validation set included 98 patients, comprised of 69 survivors and 29 fatalities, with a case fatality rate of 29.6%; 61.2% were women. Data from other hospitals (except study center) were used for external validation.

SUMMARY:
To enable emergency physicians to make well-informed triage and treatment decisions, accurate tools to evaluate the severity of diquat poisoning are needed. This study establishes severity indices for diquat poisoning (SIDPs) in assessing the risk of death for patients with acute diquat poisoning for triage purposes and 28-day mortality.

DETAILED DESCRIPTION:
Self-poisoning with pesticides is a global public health concern, and its effective control is of importance in reducing both morbidity and mortality. In China, poisoning consistently ranked as the fifth leading cause of death from 2009 to 2013, and the overall incidence rate was 39.43/100,000 population in 2019, with intentional poisoning, mostly related to self-harm. Paraquat (1,1'-dimethyl-4,4'-bipyridinium) and, after its ban in China, diquat (1,1'-ethylene-2, 2'-bipyridinium) are the agents with the highest rate of mortality due to their inherent toxicity affecting various organs paired with a lack of effective treatments. As reported from different hospitals, the inhospital case fatality rate of diquat poisoning was 18.6%, whereas the proportion of case fatalities increased to 60% after follow-up in China. Although uncommon, diquat poisoning occurs in many countries, including the United States, where 2,128 cases were identified between 1998 and 2011, and 466 cases were documented in 2023, according to the Annual Report of the National Poison Data System. The lethality of diquat underscores the necessity for precise prognosis. Estimating survival probability empowers physicians to tailor treatment decisions for patients and enhance communication, especially given the variability in capability of emergency departments (EDs) around the world.

ELIGIBILITY:
The following criteria were used for patient inclusion:

1. history of oral exposure to diquat solution reported by patient or proxy;
2. a specimen for the diquat plasma concentration collected immediately upon admission;
3. documentation that patients or, in case of unconsciousness of the patient, legal proxies were aware of and agreed to treatment plans.

Patients were excluded if:

1. they had ingested other toxicants in addition to diquat;
2. diquat was not detected in biological samples;
3. patients with over half of incomplete information;
4. patients with an exposure time (time from exposure to presentation at ED) longer than 48 hours.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute diquat poisoning
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
28-day survival | 28 days from the index date
  The primary outcome measure includes 28-day survival (survived or died).
Time from exposure to death | 28 days from the index date
  The primary outcome included time from exposure to death.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, MD, PhD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao ZX, Zhao Y, Gao J, Feng SY, Wu CP, Zhai YZ, Zhang M, Nie S, Li Y. Comparison of severity index and plasma paraquat concentration for predicting survival after paraquat poisoning: A meta-analysis. Medicine (Baltimore). 2020 Feb;99(6):e19063. doi: 10.1097/MD.0000000000019063. PMID 32028427
- [Background] Kim DS, Kang C, Kim DH, Kim SC, Lee SH, Jeong JH, Kang TS, Jung SM, Lee SB, Lee KW, Kim RB. External validation of the prognostic index in acute paraquat poisoning. Hum Exp Toxicol. 2016 Apr;35(4):366-70. doi: 10.1177/0960327115586821. Epub 2015 May 13. PMID 25977258
- [Background] Chen CK, Chen YC, Megarbane B, Yeh YT, Chaou CH, Chang CH, Lin CC. The acute paraquat poisoning mortality (APPM) score to predict the risk of death in paraquat-poisoned patients. Clin Toxicol (Phila). 2022 Apr;60(4):446-450. doi: 10.1080/15563650.2021.1979234. Epub 2021 Sep 20. PMID 34543159
- [Background] Xu S, Hu H, Jiang Z, Tang S, Zhou Y, Sheng J, Chen J, Cao Y. APACHE score, Severity Index of Paraquat Poisoning, and serum lactic acid concentration in the prognosis of paraquat poisoning of Chinese Patients. Pediatr Emerg Care. 2015 Feb;31(2):117-21. doi: 10.1097/PEC.0000000000000351. PMID 25654678
- [Background] Du Y, Mou Y. [Predictive value of 3 methods in severity evaluation and prognosis of acute paraquat poisoning]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2013 Jul;38(7):737-42. doi: 10.3969/j.issn.1672-7347.2013.07.014. Chinese. PMID 23908083
- [Background] Xing J, Chu Z, Han D, Jiang X, Zang X, Liu Y, Gao S, Sun L. Lethal diquat poisoning manifesting as central pontine myelinolysis and acute kidney injury: A case report and literature review. J Int Med Res. 2020 Jul;48(7):300060520943824. doi: 10.1177/0300060520943824. PMID 32734801
- [Background] Magalhaes N, Carvalho F, Dinis-Oliveira RJ. Human and experimental toxicology of diquat poisoning: Toxicokinetics, mechanisms of toxicity, clinical features, and treatment. Hum Exp Toxicol. 2018 Nov;37(11):1131-1160. doi: 10.1177/0960327118765330. Epub 2018 Mar 23. PMID 29569487
- [Background] Oreopoulos DG, McEvoy J. Diquat poisoning. Postgrad Med J. 1969 Sep;45(527):635-7. doi: 10.1136/pgmj.45.527.635. No abstract available. PMID 5809561
- [Background] Cai XL, Teng F, Yu X, Liu LL, Li GQ. [Four cases of acute diquat poisoning with prominent epileptoid seizure and literature review]. Zhonghua Lao Dong Wei Sheng Zhi Ye Bing Za Zhi. 2021 May 20;39(5):359-362. doi: 10.3760/cma.j.cn121094-20200224-00078. Chinese. PMID 34074081
- [Background] Yuan G, Li R, Zhao Q, Kong X, Wang Y, Wang X, Guo R. Simultaneous determination of paraquat and diquat in human plasma by HPLC-DAD: Its application in acute poisoning patients induced by these two herbicides. J Clin Lab Anal. 2021 Mar;35(3):e23669. doi: 10.1002/jcla.23669. Epub 2020 Dec 9. PMID 33296104
- [Background] Jones GM, Vale JA. Mechanisms of toxicity, clinical features, and management of diquat poisoning: a review. J Toxicol Clin Toxicol. 2000;38(2):123-8. doi: 10.1081/clt-100100926. PMID 10778908
- [Background] Saeed SA, Wilks MF, Coupe M. Acute diquat poisoning with intracerebral bleeding. Postgrad Med J. 2001 May;77(907):329-32. doi: 10.1136/pmj.77.907.329. PMID 11320278
- [Background] Huang Y, Zhang R, Meng M, Chen D, Deng Y. High-dose diquat poisoning: a case report. J Int Med Res. 2021 Jun;49(6):3000605211026117. doi: 10.1177/03000605211026117. PMID 34182818